CLINICAL TRIAL: NCT01688752
Title: Cardiometabolic Status in Childhood Acute Lymphoblastic Leukemia, A Pilot Study
Brief Title: Cardiometabolic Status in Childhood Acute Lymphoblastic Leukemia
Status: Withdrawn | Type: Observational
Why Stopped: Funding unavailable
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2012NTLS086
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood samples will be obtained for lipids (total cholesterol, triglycerides, LDL- cholesterol, HDL-cholesterol) insulin, glucose, inflammatory cytokines (CRP, IL-6, oxidized LDL), leptin, adiponectin, insulin-like growth factor 1 (IGF-1), thyroid, and gonadal function.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sibling Controls: Healthy siblings of acute lymphoblastic leukemia (ALL) subjects frequency matched by age and sex.
- Acute Lymphoblastic Leukemia Survivors: Survivors of acute lymphoblastic leukemia (ALL) who recently completed therapy.

SUMMARY:
This is a prospective cohort study assessing measures of cardiometabolic status, body composition, IR and GH response to stimulation after therapy in children (age 7-21 years) treated for ALL. Patients and sibling controls will be recruited from the Pediatric Hematology-Oncology Clinic at the University of Minnesota Amplatz Children's Hospital.

DETAILED DESCRIPTION:
This is a prospective cohort study with two groups: survivors of acute lymphoblastic leukemia (ALL) who have recently completed therapy (cases) and healthy siblings (controls) frequency matched by age and sex. Subjects in each group will have two visits. For cases, the first visit will be approximately 6 months after completion of treatment for ALL; for their siblings, the first visit occur at approximately the same time. For both cases and controls, the second visit will be 2 to 2.5 years after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Age 7 years to less than or equal to 21 years at time of study enrollment.
  * Acute lymphoblastic leukemia (ALL) as first cancer diagnosis and in first complete remission. Any subtype is eligible.
  * Study enrollment must take place at/after six months of completion of all chemotherapy.
  * Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age.
  * Any prior ALL therapy is allowable.
* Siblings

  * Age 7 years to less than or equal to 21 years at time of study enrollment.
  * Sibling of ALL patient.

Exclusion Criteria:

* Patients

  * Diagnosis of diabetes mellitus prior to ALL diagnosis or at time of study enrollment.
  * Current pregnancy
  * Prior hematopoietic cell transplant.
  * Receiving growth hormone replacement or corticosteroids at the time of enrollment.
* Siblings

  * Previously diagnosed with malignancy.
  * Diagnosis of diabetes mellitus.
  * Current pregnancy
  * Receiving growth hormone replacement or corticosteroids at the time of enrollment.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study entry is open to patients regardless of gender or ethnic background. While there will be every effort to seek out and include females and minority patients, the patient population is expected to be no different than the general pediatric oncology population seen at the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic Profile | up to 2.5-3 Years
  To determine the cardiometabolic profile (as measured by a single score based on adiposity, serum lipids, and vascular function) shortly after therapy (6 months after completion of therapy [Visit 1]) and again 2.5-3 yrs after completion of therapy (Visit 2) in 300 ALL patients, and compare with 200 sibling controls.

SECONDARY OUTCOMES:
Prevalence of Blunted Stimulated Growth Hormone Response | Between 2.5 and 3 Years
  To determine the prevalence of blunted stimulated GH response suggesting GH deficiency (peak GH <7mcg/L) in ALL survivors and controls: GH level will be obtained at baseline, then +30, +60, +90 and +120 minutes after clonidine (5 mcg/kg up to 200 mcg by mouth), followed by infusion of arginine (0.5 grams/kg up to 30 grams) with a series of GH levels at +140, +160, +180, +210, and +240 minutes. Blunted response to GH stimulation will be defined as peak GH level<7 mcg/L.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Steinberger, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota